CLINICAL TRIAL: NCT01378624
Title: Ex Vivo Effect of Fragments and Modified Forms of Surfactant Protein D on Pulmonary Immune Cells Derived From Bronchoalveolar Lavage After Segmental Allergen Challenge in Patients With Asthma and Pilot Study to Assess Local Inflammation Induced by Segmental Allergen Challenge by Magnetic Resonance Imaging
Brief Title: Ex Vivo Effect of Surfactant Protein D on Pulmonary Cells in Patients With Asthma and Pilot Study to Assess Local Inflammation Induced by Segmental Allergen Challenge by Magnetic Resonance Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Collaborators: Hannover Medical School (Other)
Responsible Party: Prof. Dr. Jens Hohlfeld, Fraunhofer ITEM
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10-07 ZAP2
Record Dates: First submitted 2011-06-17; First posted 2011-06-22 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Mild Intermittent Asthma (Gina 1)
MeSH Terms: interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bronchoscopy (Experimental)
  Interventions: Other: Bronchoscopy

INTERVENTIONS:
Other: Bronchoscopy — In brief, during the first bronchoscopy a baseline BAL and baseline endobronchial brush and forceps biopsies will be obtained and allergen as well as saline (control segment) will be instilled.
  The subjects will undergo a second bronchoscopy in order to obtain BAL from the allergen challenged segments and the saline challenged segment, and endobronchial forceps biopsies.

SUMMARY:
Ex vivo effect of fragments and modified forms of surfactant protein D on pulmonary immune cells derived from bronchoalveolar lavage after segmental allergen challenge in patients with asthma and pilot study to assess local inflammation induced by segmental allergen challenge by magnetic resonance imaging.

DETAILED DESCRIPTION:
The effect of surfactant protein D under native and altered conditions will be investigated in immune cells that are derived from bronchoalveolar lavage in patients with allergic asthma following segmental allergen challenge. The goal of this study is to elucidate the pro- versus anti-inflammatory function of SP-D molecules and to identify motifs of SP-D that have treatment potential in allergic asthma and to assess local inflammation induced by segmental allergen challenge by magnetic resonance imaging.

In addition to the patients with allergic asthma a subgroup of five healthy subjects will be included into the study to elucidate the specificity of the SP-D (surfactant protein-D) effect on the allergic inflammation in the invitro models.

The primary objective of this study is to isolate BAL cells for different invitro experiments and to assess local inflammation after segmental allergen challenge by MRI in response to the applied allergen dose.

Therefore, following a baseline BAL, allergen (2× individual dose, 1× one tenth of individual dose) and saline (1×) will be instilled into four different lung segments during a first bronchoscopy. After 24 hours during a second bronchoscopy BAL will be collected in these challenged segments to harvest invaded cells for invitro experimentation. In addition, bronchial biopsies and epithelial brushes will be taken to assess the degree of local inflammation in bronchial mucosa and to study the activation of airway epithelium following allergen challenge.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written informed consent
* Physician diagnosis of mild asthma according to GINA guidelines (1;7)
* Nonsmokers with a history of less than 1 pack a year having been nonsmokers for at least the last five years
* FEV1 80% of predicted
* Positive skin prick test for grass mix or D. pteronyssinus at or within 12 months prior to the screening visit
* Positive response to an incremental inhaled allergen challenge with house dust mite allergen or grass pollen allergen
* Women will be considered for inclusion if they are:

  * Not pregnant, as confirmed by pregnancy test, and not nursing
  * Of non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is pre-menarchial or post-menopausal, with documented proof of hysterectomy or tubal ligation, or meet clinical criteria for menopause and has been amenorrhoeic for more than 1 year prior to the screening visit)o of childbearing potential and using a highly effective method of contraception during the entire study (vasectomized partner, sexual abstinence
  * The lifestyle of the female should be such that there is complete abstinence from intercourse from two weeks prior to the study until at least 72 hours after the end of the study
  * Implants, injectables, combined oral contraceptives, hormonal IUDs, or double barrier methods (i.e. any double combination of IUD, condom with spermicidal gel,diaphragm, sponge, and cervical cap)

Exclusion Criteria:

* History of upper or lower respiratory tract infection four weeks prior to the informed consent visit
* Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, psychiatric disease, endocrine disease, infectious disease, inflammatory disease, or pulmonary disease (including but not confined to chronic bronchitis, emphysema, tuberculosis, bronchiectasis or cystic fibrosis).
* Clinically significant pathological findings in safety laboratory tests
* Regular intake of any medication other than short acting inhaled beta agonists, paracetamol for pain relief, birth control medication, hormonal replacement therapy, dietary and vitamin supplements
* Specific Immunotherapy (SIT) within two years prior to the study
* Use of anti-inflammatory medication including systemic or inhaled corticosteroid within the last four weeks
* Any history of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnea, respiratory arrest or hypoxic seizures.
* Suspected hypersensitivity to any ingredients of the medication in line with bronchoscopy (bronchodilators, sedatives and local anesthetics)
* Conditions or factors, which would make the subject unlikely to be able to undergo bronchoscopy or incremental allergen challenge
* Conditions or factors, which would make the subject unable to undergo MRI such as metal containing implants, remainders of shell splinters or bullets, or claustrophobia.
* History of drug or alcohol abuse
* Suspected inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study.
* Participation in a clinical trial 30 days prior to enrollment
* Segmental allergen challenge three months prior to treatment
* Risk of non-compliance with study procedures
* Calculated GFR <30 ml/min/1.73 m2
* Known allergy to MRI based contrast agents
* Donation of more than 500 ml of blood in the preceding 9 weeks before the trial examination
* Hb Hemoglobin below lower limit of normal value

Additional Inclusion Criteria for healthy control subjects:

* Healthy subjects with no clinical evidence of allergic rhinitis and respiratory disease (e.g. asthma)
* Negative skin prick test for grass mix or D. pteronyssinus at or within 12 months prior to the screening visit
* Negative response to an incremental metacholine challenge (PC20 ≥ 8mg/ml)
* Total IgE (Immunglobulin E) <100 IU/ml

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2011-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change in local inflammation | Baseline, 6 and 24 hours post segmental allergen challenge
  Magnetic resonance imaging to assess local inflammation prior to as well as 6 h and 24 h after segmental allergen challenge
Change of numbers of matured dendritic cells | Baseline and 24 h post segmental allergen challenge
  Change of numbers of matured dendritic cells in vitro in the absence and presence of surfactant protein D.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hohlfeld, MD, Professor, Principal Investigator — Fraunhofer ITEM
Locations (1):
- Fraunhofer ITEM, Hanover, Lower Saxony, Germany